CLINICAL TRIAL: NCT06761859
Title: The Effect of Aromatherapy Inhalation on the Therapeutic Relationship and Work Stress Levels of Psychiatric Nurses
Brief Title: Aromatherapy Inhalation in Psychiatric Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SERDAR TÜRKYILMAZ (Other Government)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Sponsor-Investigator, SERDAR TÜRKYILMAZ, Nurse, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0009-0003-2884-5320
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Aromatherapy
Keywords: Psychiatric nursing; inhalation; aromatherapy; therapeutic relationship; work stress
MeSH Terms: conditions — Respiratory Aspiration; Occupational Stress | interventions — Psychiatric Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In this study, aromatherapy inhalation will be applied to psychiatric nurses in the experimental group. Aromatherapy inhalation using 2% diluted lavender essential oil will be applied to 33 psychiatric nurses in the experimental group, 30 minutes before starting work, every other day during a week. The "General Job Stress Scale (GJSS)" and "Therapeutic Relationship Evaluation Scale-Nurse Form (TRES-NF)" inventories will be filled out by 33 psychiatric nurses in the experimental group before and after aromatherapy inhalation, and by 33 psychiatric nurses in the control group simultaneously with the psychiatric nurses in the experimental group.
  Interventions: Other: Aromatherapy Inhalation in Psychiatric Nurses
- Control group (No Intervention): There will be no training or intervention. No intervention will be made to the 33 psychiatric nurses in the control group. The psychiatric nurses in the control group will be asked to fill out the "General Job Stress Scale (GJSS)" and "Therapeutic Relationship Evaluation Scale-Nurse Form (TRES-NF)" inventories simultaneously with the 33 psychiatric nurses in the experimental group.

INTERVENTIONS:
Other: Aromatherapy Inhalation in Psychiatric Nurses — Aromatherapy inhalation using 2% diluted lavender essential oil will be applied to 33 psychiatric nurses in the experimental group, 30 minutes before starting work, every other day during a week. The lavender essential oil to be used in the study will be dropped 3 drops onto a cotton handkerchief cut into a disc shape and fixed to the clothes of the psychiatric nurses, 20 cm away from their noses, and they will be asked to inhale it for 30 minutes.
  Arms: Experimental group

SUMMARY:
In this study will be conducted with a total of 66 psychiatric nurses who meet the inclusion and exclusion criteria and are working at Ankara Etlik City Hospital Psychiatry Clinic between January 1, 2025 and March 31, 2025.

DETAILED DESCRIPTION:
In this study, aromatherapy inhalation will be applied to psychiatric nurses in the experimental group. Aromatherapy inhalation using 2% diluted lavender essential oil will be applied to 33 psychiatric nurses in the experimental group, 30 minutes before starting work, every other day during a week. The "General Job Stress Scale (GJSS)" and "Therapeutic Relationship Evaluation Scale-Nurse Form (TRES-NF)" inventories will be filled out by 33 psychiatric nurses in the experimental group before and after aromatherapy inhalation, and by 33 psychiatric nurses in the control group simultaneously with the psychiatric nurses in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Written permission was obtained before participating in the study
* Having worked in the psychiatry departments of the relevant institution for at least 1 year
* Working in the psychiatry departments of the relevant institution during the study dates
* Not sensitive to the odor of lavender essential oil

Exclusion Criteria:

* Previous experience with aromatherapy
* Sensitivity and allergy to lavender essential oil
* Willingly leaving the study while the study was ongoing
* Leaving the job during the study period
* General condition changes during the study period (developing allergies, getting sick, taking annual leave, taking leave with a health report)
* Becoming a service responsible nurse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
General Job Stress Scale (GJSS) | Change from before implementation, after practice is completed (1th week)
  The Turkish validity and reliability of the scale developed by De Bruin (2006) to measure the general job stress of employees was provided by Teleş (2020). The scale has a one-dimensional structure that addresses the emotional, cognitive, motivational and social consequences of job stress. The scale, which has no sub-dimensions and consists of a five-point Likert-type and nine items, is stated as "1=Never, 2=Rarely, 3=Sometimes, 4=Mostly, 5=Always". The total score to be obtained from the scale is a concrete expression of job stress and a high score to be obtained from the scale indicates that high job stress is experienced. As a result of the validity and reliability study conducted by Teleş (2020), the Cronbach alpha coefficient of the scale was stated as 0.91 (De Bruin, 2006; Teleş, 2020).
Therapeutic Relationship Evaluation Scale-Nurse Form (TRES-NF) | Change from before implementation, after practice is completed (1th week)
  Developed by Coelho et al. (2021) to assess the quality of the therapeutic relationship between psychiatric nurses and psychiatric patients, the Turkish validity and reliability of the scale was established by Duran and Polat (2023). The scale, which consists of a five-point Likert type and 25 items, can be used in one dimension or with four subdimensions as "empathy, self-awareness, participation in care, and orientation". The answers to each item in the scale are specified as "1=Never, 2=Rarely, 3=Sometimes, 4=Frequently, 5=Always". It has been stated that a minimum of 25 and a maximum of 125 points can be obtained if the scale is used in one dimension. It has been stated that if the scale is used in other subdimensions, 5-25 points can be obtained from the empathy subdimension, 6-30 from the self-awareness subdimension, 8-40 from the participation in care subdimension, and 6-30 from the orientation subdimension. As a result of their validity and reliability study, Duran and Polat (

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided